CLINICAL TRIAL: NCT02451683
Title: Corticospinal Function After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Monica Perez, Scientific Chair Arms + Hands AbilityLab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00210458; R01NS090622-01 (NIH)
Record Dates: First submitted 2015-05-11; First posted 2015-05-22 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injury
Keywords: SCI
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electrophysiology Assessment of Time Domain (Other): Assessment of electrophysiology in the time domain to examin temporal organization of corticospinal function
  Interventions: Other: Electrophysiology Assessment of Time Domain; Other: Training with some stimulation
- Electrophysiology Assessment of Location (Experimental): Assessment of electrophysiology to examine spatial organization of corticospinal function
  Interventions: Other: Electrophysiology Assessment of Location; Other: Training with some stimulation
- Training with some stimulation (Active Comparator): Training with non-invasive stimulation and training with sham stimulation
  Interventions: Other: Training with some stimulation

INTERVENTIONS:
Other: Electrophysiology Assessment of Time Domain — Kinematics, Spinal Cord Excitability and Cortical Spinal Motor Excitability.
  Arms: Electrophysiology Assessment of Time Domain
Other: Electrophysiology Assessment of Location — Kinematics, Spinal Cord Excitability and Cortical Spinal Motor Excitability
  Arms: Electrophysiology Assessment of Location
Other: Training with some stimulation — motor task combined with real or sham stimulation

SUMMARY:
The investigator's overall goal is to develop new strategies to test optimization of Spike-timing-dependent plasticity (STDP) doses to maximize strategy to restore upper and lower-limb motor function in individuals with spinal cord injury (SCI). The investigator proposes to use modern electrophysiological methods to enhance the efficacy of residual corticospinal connections. Defining the neural basis by which corticospinal volleys generate muscle responses will provide crucial information required to maximize residual motor output. The investigator's specific goals are to: 1) determine the temporal and spatial organization of corticospinal volleys and motor cortical representations of upper-limb muscles after incomplete cervical SCI and 2) develop methodologies to promote recovery of function. The investigator's focus on reach and grasp movements because of their importance in daily life activities.

DETAILED DESCRIPTION:
This study will determine the temporal organization of corticospinal volleys during reach and grasp movements. Multiple descending volleys in the corticospinal tract generate multiple peaks in muscle responses (indirect (I)-waves). I-waves are a mechanism by which corticospinal neurons are transynaptically activated at periodic intervals of ~1.5 ms. This periodic activation contributes to the recruitment of spinal motoneurons and generation of movement. we will use paired-TMS to examine I-waves in surface EMG recordings from upper-limb muscles during reach and grasp movements.

We will also identify motor cortical maps of upper-limb muscles involved in reach and grasp movements. We will use TMS guided by a frameless neuronavigation system to define the size and location of motor cortical maps of upper-limb muscles during reach and grasp movements. We will be able to determine overlaps and functional interactions between distal and proximal arm motor cortical representations. Our preliminary data shows that finger and biceps cortical maps largely overlap during reach and grasp movements in controls but considerable less in patients

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for individuals with SCI:

  1. Male and females between 18-85 years,
  2. Chronic SCI (≥ 6 months post injury),
  3. Cervical injury at C8 or above,
  4. Intact or impaired but not absent innervations in dermatomes C6, C7, and C8 using the American Spinal Injury Association sensory scores, and
  5. Ability to reach and grasp a small object located at least 8 cm forward, above, and laterally without leaning forward with the trunk

Inclusion criteria for healthy controls:

1. Male and females between 18-85 years,
2. Right handed,
3. Ability to reach and grasp a small object located at least 8 cm forward, above, and laterally without leaning forward with the trunk

Exclusion Criteria:

* Exclusion criteria for individuals with SCI and Healthy Controls:

  1. Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
  2. Any debilitating disease prior to the SCI that caused exercise intolerance
  3. Premorbid, ongoing major depression or psychosis, altered cognitive status
  4. History of head injury or stroke
  5. Pacemaker
  6. Metal plate in skull
  7. History of seizures
  8. Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants
  9. Pregnant females
  10. Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida or herniated cervical disk.
  11. History of brain tumor and or brain infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Upper-limb motor function | 5 months
  measured by functional tests of hand/arm motor function

SECONDARY OUTCOMES:
Cortical Neurophysiological Outcome | 5 months
  measured by the maps area and overlap in millimeters
Change in Sensorimotor Function | 5 months
  measured by upper-limb movements scale from 1(dependent) to 7 (independent).

CONTACTS AND LOCATIONS:
Overall Officials: Monica Perez, PT PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No